CLINICAL TRIAL: NCT06066827
Title: Hair Regeneration in Androgenetic Alopecia Using Secretome of Adipose-derived Stem Cells (ADSC) and Minoxidil: A Comparative Study of Three Groups
Brief Title: Hair Regeneration in Androgenetic Alopecia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. dr. Lili Legiawati, SpKK(K) (Other)
Collaborators: Ministry of Education, Culture, Research, and Technology, Republic of Indonesia (Unknown); PT. Kimia Farma (Persero) Tbk (Industry)
Responsible Party: Sponsor-Investigator, Dr. dr. Lili Legiawati, SpKK(K), Principal Investigator, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 977/UN2.F1/ETIK/PPM.00.02/2023
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Androgenetic Alopecia
Keywords: Secretome; Minoxidil; Skin; Androgenetic alopecia
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Intervention Model Description: Each subject will receive an injection of the secretome from ADCS's, topical minoxidil, or both.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This study was a single-blind clinical trial, masking the investigator and outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Minoxidil (Experimental): The drug used is minoxidil 5% solutions for topical use, 1 cc, 2 times a day, every day for 12 weeks
  Interventions: Drug: Minoxidil Topical
- Secretome from Adipose-Derived Stem Cells (Experimental): Secretom concentrate of Adipose-Derived Stem Cells (ADSCs) 2cc, injected to the scalp on weeks 0, 4, and 8 of the study
  Interventions: Other: Secretome from adipose-derived stem cells
- Minoxidil + Secretome (Experimental): The subject received both minoxidil and secretome from ADSCs, with the same dosage form, dosage, frequency, and duration
  Interventions: Combination Product: Combination of minoxidil and secretome from adipose-derived stem cells

INTERVENTIONS:
Drug: Minoxidil Topical — 20 subjects received minoxidil only for the treatment of AGA
  Arms: Minoxidil
Other: Secretome from adipose-derived stem cells — 20 subjects received the injection of secretome from adipose-derived stem cells only for the treatment of AGA
  Arms: Secretome from Adipose-Derived Stem Cells
Combination Product: Combination of minoxidil and secretome from adipose-derived stem cells — 20 subjects received both minoxidil and injection of secretome from adipose-derived stem cells for the treatment of AGA
  Arms: Minoxidil + Secretome

SUMMARY:
This clinical trial study aims to compare the effectiveness and safety of secretome from ADSCs with minoxidil in AGA cases, to provide future reference or standard in the application of cell-based therapy and its derivatives in AGA cases. The subject of this study is androgenetic alopecia population. The main questions it aims to answer are:

* Is the secretome of ADSC's effective compared to minoxidil?
* Is the secretome of ADSC's safe compared to minoxidil?
* Is the combination of the secretome of ADSC's and minoxidil better in safety and effectiveness compared to secretome or minoxidil alone?

DETAILED DESCRIPTION:
This study was a single-blind clinical trial using an experimental research design on subjects with androgenetic alopecia. Variables tested in this study were the method of "treatment of AGA by administering secretome concentrate alone, compared to using minoxidil alone and with a combination of both."

Subjects were divided into 3 groups:

* 20 subjects received secretome
* 20 subjects received minoxidil
* 20 subjects received both treatments Participants will undergo history taking, and a physical examination (including vital signs, body weight, and hair pull test). Pictures of patients' head were then taken and the hair loss degree was graded using Hamilton-Norwood. Hair growth was evaluated every month starting from months 0, 1, 2, and 3. Clinical assessment of hair growth was examined through physical and supporting examinations including photography, trichoscan, and trichoscopy.

The sample size for this study was calculated with the help of G*Power version 3.1 software (Heinrich-Heine-Universität Düsseldorf, Düsseldorf, Germany).

The inclusion and exclusion criteria are applied. Statistical data were analyzed using SPSS® version 21 software. On numerical data, normality analysis was carried out using the Kolmogorov-Smirnov test.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18-59 years
* Clinical presentation of AGA with Hamilton-Norwood Grade III-VI
* Willing to be a research subject, sign a consent form, and commit to regular follow-up visits

Exclusion Criteria:

* Hair loss other than AGA, including telogen effluvium, alopecia areata, trichotillomania, secondary syphilis, systemic lupus erythematosus hair loss due to chemotherapy, autoimmune conditions, or malignancies.
* Patients taking oral medications or vitamins aimed at increasing hair growth in the last month
* Patients applying topical medications aimed at increasing hair growth in the last 2 weeks
* Patients with active bacterial, viral, or fungal infections on the scalp
* Patients undergoing AGA therapy cosmetic procedures in the form of PRP injections, laser procedures, or micro-needling in the last 3 months

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of alopecia in physical examination | Week 0 (baseline), week 4 after intervention, week 8 after intervention, week 12 (end of trial)
  The investigator conduct a scalp examination every 4 weeks until the twelfth week to measure the improvement of alopecia with Hamilton-Norwood scale
Macroscopic hair growth documented | Week 0 (baseline), week 4 after intervention, week 8 after intervention, week 12 (end of trial)
  The investigator conducted documentation of the subject in 7 positions, so that the improvement of alopecia can be seen from various directions
Microscopic hair growth evaluated by Trichoscopy | Week 0 (baseline), week 4 after intervention, week 8 after intervention, week 12 (end of trial)
  Microscopic hair growth was documented using Heine® Delta 20 Plus (Heine, Germany) dermoscopy for qualitative measurement
Microscopic hair growth evaluated by Trichoscan | Week 0 (baseline), week 4 after intervention, week 8 after intervention, week 12 (end of trial)
  The investigator use Fotofinder® medicam 1000 s video-trichoscopy (FotoFinder Systems GmbH, Germany) for quantitative measurements, such as hair rate anagen (%), hair rate telogen (%), hair rate terminal (%), and hair rate vellus (%)

SECONDARY OUTCOMES:
Patient satisfaction | Week 12 (end of trial)
  The patient satisfaction scale using a linear analog scale with a scale of 1-7 (1 = no result, 7 = very satisfactory outcome) and was evaluated at the last treatment session.

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - RSUP Nasional Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta
  - Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Legiawati L, Sitohang IBS, Yusharyahya SN, Sirait SP, Novianto E, Liem IK, Kurniawati T, Putri IS, Rahmadika FD, Hakiki NP, Lauren BC. Hair regeneration in androgenetic alopecia using secretome of adipose-derived stem cells (ADSC) and minoxidil: a comparative study of three groups. Arch Dermatol Res. 2025 Mar 1;317(1):486. doi: 10.1007/s00403-025-04006-3. PMID 40021536